CLINICAL TRIAL: NCT01171898
Title: An Open-Label, Phase 1/2, Safety, Pharmacokinetic and Proof-of-Concept Study of ARN-509 in Patients With Progressive Advanced Castration-Resistant Prostate Cancer
Brief Title: Safety, Pharmacokinetic and Proof-of-Concept Study of ARN-509 (Apalutamide) in Castration-Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103304; ARN-509-001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Non-Metastatic; Rising PSA; Castration-Resistant; Treatment-Naive; Post-abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Escalation Cohort (Phase 1) (Experimental): ARN-509 will be administered at a starting dose of 30 milligram per day (mg/day), with escalations to 60 mg, 90 mg, 120 mg, 180 mg, 240 mg, 300 mg, 390 mg, and 480 mg daily. Once Recommended Phase 2 Dose (RP2D) has been selected, Phase 1 participants being treated at the lower dose levels will be allowed to escalate to the RP2D level at the discretion of the primary investigator.
  Interventions: Drug: ARN-509 (Phase 1)
- Non-metastatic CRPC (Phase 2) (Experimental): Participants with non-metastatic, treatment-naive Castration-Resistant Prostate Cancer (CRPC) with rapidly rising Prostate Specific Antigen (PSA) will be enrolled. ARN-509 will be administered at Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D), determined in Phase 1.
  Interventions: Drug: ARN-509 (Phase 2)
- Treatment-naive metastatic CRPC (Phase 2) (Experimental): Participants with treatment-naive metastatic CRPC will be enrolled. ARN-509 will be administered at MTD and/or RP2D, determined in Phase 1.
  Interventions: Drug: ARN-509 (Phase 2)
- Post-abiraterone metastatic CRPC (Phase 2) (Experimental): Participants with metastatic CRPC that are chemotherapy-naive, but have been previously treated with abiraterone will be enrolled. ARN-509 will be administered at MTD and/or RP2D, determined in Phase 1.
  Interventions: Drug: ARN-509 (Phase 2)

INTERVENTIONS:
Drug: ARN-509 (Phase 1) — ARN-509 will be administered at a starting dose of 30 milligram per day (mg/day), with escalations to 60 mg, 90 mg, 120 mg, 180 mg, 240 mg, 300 mg, 390 mg, and 480 mg daily.
  Arms: Dose Escalation Cohort (Phase 1)
Drug: ARN-509 (Phase 2) — ARN-509 will be administered at Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D), determined in Phase 1.
  Arms: Non-metastatic CRPC (Phase 2); Post-abiraterone metastatic CRPC (Phase 2); Treatment-naive metastatic CRPC (Phase 2)

SUMMARY:
The purpose of this study is to assess the safety and activity of ARN-509 in men with advanced castration resistant prostate cancer. Patients will first be enrolled into Phase 1 of the study to identify a tolerable dose for the Phase 2 portion of the study. In the Phase 2, 3 different cohorts of patients will be enrolled to evaluate the safety and activity of ARN-509.

ELIGIBILITY:
NON-METASTATIC CRPC

Inclusion Criteria

1. Histologically or cytologically proven prostate cancer with high risk for development of metastases, defined as either a PSA value >=8 ng/mL within the last 3 months or PSA Doubling Time <=10 months
2. Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration)
3. Castrate levels of serum testosterone of less than or equal to 50 ng/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. A life expectancy of at least 3 months

Exclusion Criteria

1. Distant metastases, including CNS and vertebral or meningeal involvement
2. Prior treatment with MDV3100
3. Prior treatment with abiraterone
4. Prior treatment with ketoconazole
5. Concurrent treatment with medications known to have seizure potential
6. Concurrent treatment with corticosteroids. If they are already on steroids, patients will be allowed to enroll on the study but will need to taper off as soon as possible.
7. QTc > 450 msec
8. History of seizure or condition that may predispose to seizure
9. Evidence of severe or uncontrolled systemic disease or HIV infection

METASTATIC CRPC, TREATMENT-NAIVE

Inclusion Criteria

1. Histologically or cytologically proven prostate cancer with progressive disease based on either PSA or radiographic progression
2. Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration)
3. Castrate levels of serum testosterone of less than or equal to 50 ng/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. A life expectancy of at least 3 months

Exclusion Criteria

1. History of, or current metastases in the brain or untreated spinal cord compression
2. Prior treatment with MDV3100
3. Prior treatment with abiraterone
4. Prior treatment with ketoconazole
5. Concurrent treatment with medications known to have seizure potential
6. Concurrent treatment with corticosteroids. If they are already on steroids, patients will be allowed to enroll on the study but will need to taper off as soon as possible.
7. QTc > 450 msec
8. History of seizure or condition that may predispose to seizure
9. Evidence of severe or uncontrolled systemic disease or HIV infection

METASTATIC CRPC, CHEMOTHERAPY-NAIVE, POST-ABIRATERONE

Inclusion Criteria

1. Histologically or cytologically proven prostate cancer with progressive disease based on either PSA or radiographic progression
2. Ongoing androgen depletion therapy with a Gonadotropin Releasing Hormone (GnRH) analogue or inhibitor, or orchiectomy (i.e., surgical or medical castration)
3. Castrate levels of serum testosterone of less than or equal to 50 ng/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. A life expectancy of at least 3 months
6. Patients must have received a minimum of 6 months of abiraterone treatment prior to disease progression

Exclusion Criteria

1. History of, or current metastases in the brain or untreated spinal cord compression
2. Prior treatment with MDV3100
3. Prior treatment with ketoconazole
4. Concurrent treatment with medications known to have seizure potential
5. Concurrent treatment with corticosteroids. If they are already on steroids, patients will be allowed to enroll on the study but will need to taper off as soon as possible.
6. QTc > 450 msec
7. History of seizure or condition that may predispose to seizure
8. Evidence of severe or uncontrolled systemic disease or HIV infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-07-26 (Actual); Primary Completion 2012-08-20 (Actual); Study Completion 2025-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (15):
- United States (15):
  - San Diego, California
  - San Francisco, California
  - Atlanta, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Omaha, Nebraska
  - New York, New York
  - Raleigh, North Carolina
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Myrtle Beach, South Carolina
  - Dallas, Texas
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Rathkopf DE, Smith MR, Ryan CJ, Berry WR, Shore ND, Liu G, Higano CS, Alumkal JJ, Hauke R, Tutrone RF, Saleh M, Chow Maneval E, Thomas S, Ricci DS, Yu MK, de Boer CJ, Trinh A, Kheoh T, Bandekar R, Scher HI, Antonarakis ES. Androgen receptor mutations in patients with castration-resistant prostate cancer treated with apalutamide. Ann Oncol. 2017 Sep 1;28(9):2264-2271. doi: 10.1093/annonc/mdx283. PMID 28633425
- [Derived] Smith MR, Antonarakis ES, Ryan CJ, Berry WR, Shore ND, Liu G, Alumkal JJ, Higano CS, Chow Maneval E, Bandekar R, de Boer CJ, Yu MK, Rathkopf DE. Phase 2 Study of the Safety and Antitumor Activity of Apalutamide (ARN-509), a Potent Androgen Receptor Antagonist, in the High-risk Nonmetastatic Castration-resistant Prostate Cancer Cohort. Eur Urol. 2016 Dec;70(6):963-970. doi: 10.1016/j.eururo.2016.04.023. Epub 2016 May 6. PMID 27160947

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Cohort (Phase 1): Participants received apalutamide (ARN-509) at a starting dose of 30 milligram per day (mg/day), with escalations to 60 mg, 90 mg, 120 mg, 180 mg, 240 mg, 300 mg, 390 mg, and 480 mg daily (up to 240 mg once daily and at higher doses of 300/390/480 mg twice daily dosing). Once Recommended Phase 2 Dose (RP2D) was selected, Phase 1 participants being treated at the lower dose levels were allowed to escalate to the RP2D level (240 mg) at the discretion of the primary investigator.
- Cohort 1: Non-metastatic CRPC (Phase 2): Participants with non-metastatic, treatment naive Castration-Resistant Prostate Cancer (CRPC) with rapidly rising Prostate Specific Antigen (PSA) enrolled in Cohort 1 of Phase 2, received apalutamide at Maximum Tolerated Dose (MTD) and/or RP2D of 240 mg, determined in Phase 1.
- Cohort 2: Treatment-naive Metastatic CRPC (Phase 2): CRPC (Phase 2) Participants with metastatic CRPC who had not received chemotherapy for metastatic disease or prior abiraterone acetate (treatmentnaive) were enrolled in Cohort 2 of Phase 2, received apalutamide at MTD and/or RP2D of 240 mg, determined in Phase 1.
- Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2): Participants with metastatic CRPC that were chemotherapynaive, but had been previously treated with abiraterone acetate enrolled in Cohort 3 of Phase 2 received apalutamide at MTD and/or RP2D of 240 mg, determined in Phase 1.
Period: Overall Study
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
Started | 30 | 51 | 25 | 21
Completed | 26 | 32 | 13 | 15
Not Completed | 4 | 19 | 12 | 6
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 6 | 3
Not completed — Terminated by Sponsor | 1 | 0 | 0 | 0
Not completed — Ongoing | 1 | 9 | 3 | 0
Not completed — Other | 1 | 5 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Cohort (Phase 1): Participants received apalutamide at a starting dose of 30 milligram per day (mg/day), with escalations to 60 mg, 90 mg, 120 mg, 180 mg, 240 mg, 300 mg, 390 mg, and 480 mg daily (up to 240 mg once daily and at higher doses of 300/390/480 mg twice daily dosing). Once Recommended Phase 2 Dose (RP2D) was selected, Phase 1 participants being treated at the lower dose levels were allowed to escalate to the RP2D level (240 mg) at the discretion of the primary investigator.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2) | Total
Number analyzed (Participants) | 30 | 51 | 25 | 21 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.44) | 72.8 (8.73) | 70 (11.8) | 67.4 (9.28) | 70.2 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 30 | 51 | 25 | 21 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 29 | 49 | 25 | 21 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 2 | 5
  White | 30 | 47 | 25 | 19 | 121
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 51 | 25 | 21 | 127

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 and 2: Percentage of Participants With Greater Than or Equal to (>=) 50 Percent (%) Reduction in Prostate-Specific Antigen (PSA) at Week 12
Description: Percentage of participants with >=50% decrease in PSA compared to baseline were assessed at Week 12. PSA progression was defined by the protocol-specific Prostate Cancer Working Group 2 (PCWG2) criteria: PSA increase greater than or equal to [>=] 25 percent [%] and >=2 nanogram per milliliter [ng/mL] above the nadir confirmed >=3 weeks later; or >=25% and >=2 ng/mL above baseline PSA after 12 weeks.
Time Frame: Week 12
Population: Modified intent-to-treat (mITT) population included all participants who received at least one dose of apalutamide and who were eligible for the cohort that they were enrolled in.
Measure: Number; unit: Percentage of Participants
Groups:
- Cohort 2: Treatment-naive Metastatic CRPC (Phase 2): Participants with metastatic CRPC who had not received chemotherapy for metastatic disease or prior abiraterone acetate (treatment-naive) were enrolled in Cohort 2 of Phase 2, received apalutamide at MTD and/or RP2D of 240 mg, determined in Phase 1.
- Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2): Participants with metastatic CRPC that were chemotherapy-naive, but had been previously treated with abiraterone acetate enrolled in Cohort 3 of Phase 2 received apalutamide at MTD and/or RP2D of 240 mg, determined in Phase 1.
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
Number analyzed (Participants) | 30 | 47 | 25 | 18
Percentage of Participants | 47 | 89 | 88 | 22

2. Secondary Outcome: Phase 1 and 2: Median Time to PSA Progression
Description: Time to PSA progression was measured as the time interval from the date of the first dose to the date of PSA progression as defined by the PCWG2 criteria. PCWG2 criteria: For participants who achieved >=50% decrease from the baseline PSA, assessment of time to disease progression was when the PSA increased 25% and at a minimum of 2 ng/mL above the nadir at 3 or more weeks later. For participants without a PSA decrease, the time for progression was calculated at the time when the PSA progression was >=25% and >=2 ng/mL after 12 weeks.
Time Frame: Up to approximately 7 years
Population: mITT population included all participants who received at least one dose of apalutamide and who were eligible for the cohort that they were enrolled in.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
Number analyzed (Participants) | 30 | 47 | 25 | 18
Months | 4.9 [3.9 to 9.5] | 24.0 [16.30 to 35.0] | 16.5 [5.6 to 59.5] | 3.0 [2.7 to 4.7]

3. Secondary Outcome: Phase 2: Median Metastasis-Free Survival (MFS)
Description: MFS was defined as the time from the start of treatment until new metastatic lesions were observed on Computed Tomography/ Magnetic Resonance Imaging (CT/MRI) scans or radionuclide bone scans (according to PCWG2 criteria: appearance of >=2 new lesions, and, for the first reassessment only, a confirmatory scan performed 6 or more weeks later that showed at least 2 or more additional new lesions) or death, whichever occurred first.
Time Frame: Up to approximately 7 years
Population: mITT population included all participants who received at least 1 dose of apalutamide and were eligible for cohort that they were enrolled in. MFS results are reported for Cohort 1 (Phase 2) participants only as MFS analysis was not performed for other cohorts that is Dose Escalation Cohort (Phase 1) and Cohort 2, 3 (Phase 2) per planned analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Non-metastatic CRPC (Phase 2)
Number analyzed (Participants) | 47
Months | 21.6 [11.5 to 40.9]

4. Secondary Outcome: Phase 1 and 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the radiographic disease progression or death, whichever occurred first. Radiographic progression defined by at least one of the following: a) Soft tissue progression by modified RECIST confirmed on repeat imaging >= 6 weeks later; b) Progression by bone scans: 1) first bone scan with >= 2 new lesions compared to baseline observed <12 weeks from start date and confirmed on a second bone scan >=6 weeks later that showed >=2 additional lesions (a total of >=4 new lesions compared to baseline); or 2) first bone scan with >=2 new lesions compared to baseline observed >=12 weeks from start date and the new lesions verified on the next bone scan >=6 weeks later (a total of >=2 new lesions compared to baseline).
Time Frame: Up to approximately 7 years
Population: mITT population included all participants who received at least 1 dose of apalutamide and who were eligible for cohort that they were enrolled in. PFS results are reported for Dose Escalation Cohort (Phase 1) and cohort 2, 3 (Phase 2) as no PFS analysis was performed for Cohort 1 of Phase 2 per planned analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
Number analyzed (Participants) | 30 | 25 | 18
Months | 16.82 [11.76 to NA] — Here NA signifies that the upper limit of Confidence Interval (CI) was not estimable due to lesser number of events. | 36.37 [16.66 to NA] — Here NA signifies that the upper limit of Confidence Interval (CI) was not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower and upper limit of Confidence Interval (CI) were not estimable due to lesser number of events.

5. Secondary Outcome: Phase 1 and 2: Objective Response Rate
Description: Objective Response Rate was defined as the percentage of participants with best overall response (OR) of confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.0 (RECIST). Where, CR defined as disappearance of all target lesions. Any pathological lymph nodes must had reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of the diameters of the target lesions. Confirmed responses were those that persisted on repeat imaging study for at least 4 weeks after initial documentation of response.
Time Frame: Up to approximately 7 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
Number analyzed (Participants) | 30 | 47 | 25 | 18
Percentage of Participants | 20 [2.52 to 55.61] | 0 [0 to 97.50] | 50 [15.70 to 84.30] | 0 [0 to 30.85]

ADVERSE EVENTS:
Time Frame: Up to approximately 7 years
Description: Safety population included all participants who received at least one dose of apalutamide.
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1: Non-metastatic CRPC (Phase 2) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/51 | 2/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 7/30 | 16/51 | 10/25 | 6/21
Other Adverse Events (participants affected / at risk) | 29/30 | 49/51 | 25/25 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort (Phase 1) (N=30) | Cohort 1: Non-metastatic CRPC (Phase 2) (N=51) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) (N=25) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2) (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal Ganglia Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0
Nerve Root Compression (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder Outlet Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort (Phase 1) (N=30) | Cohort 1: Non-metastatic CRPC (Phase 2) (N=51) | Cohort 2: Treatment-naive Metastatic CRPC (Phase 2) (N=25) | Cohort 3: Post-Abiraterone Metastatic CRPC (Phase 2) (N=21)
Anaemia (Blood and lymphatic system disorders) | 3 | 9 | 5 | 3
Hypothyroidism (Endocrine disorders) | 3 | 11 | 3 | 1
Vision Blurred (Eye disorders) | 1 | 4 | 2 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 5 | 4 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 5 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 10 | 12 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 6 | 2 | 3
Constipation (Gastrointestinal disorders) | 10 | 9 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 9 | 22 | 11 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 7 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 7 | 4 | 0
Nausea (Gastrointestinal disorders) | 9 | 20 | 14 | 7
Vomiting (Gastrointestinal disorders) | 2 | 7 | 4 | 4
Asthenia (General disorders) | 1 | 6 | 1 | 1
Chest Pain (General disorders) | 2 | 2 | 3 | 2
Fatigue (General disorders) | 16 | 34 | 15 | 11
Oedema Peripheral (General disorders) | 6 | 10 | 4 | 1
Pain (General disorders) | 6 | 4 | 3 | 2
Pyrexia (General disorders) | 2 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 10 | 5 | 1
Sinusitis (Infections and infestations) | 1 | 4 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 8 | 4 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 8 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 9 | 0 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 3 | 3 | 2
Weight Decreased (Investigations) | 1 | 9 | 2 | 2
Weight Increased (Investigations) | 2 | 1 | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 7 | 4 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 5 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12 | 7 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 14 | 6 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 7 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 2 | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4 | 3
Dizziness (Nervous system disorders) | 3 | 7 | 4 | 2
Dysgeusia (Nervous system disorders) | 1 | 11 | 2 | 2
Headache (Nervous system disorders) | 6 | 8 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 1 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 3 | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 4 | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 5 | 4 | 1
Dysuria (Renal and urinary disorders) | 4 | 3 | 2 | 0
Haematuria (Renal and urinary disorders) | 4 | 7 | 2 | 2
Nocturia (Renal and urinary disorders) | 3 | 4 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 9 | 3 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 7 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 7 | 4 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 0
Hot Flush (Vascular disorders) | 5 | 10 | 5 | 0
Hypertension (Vascular disorders) | 1 | 7 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 2 | 0
Cataract (Eye disorders) | 0 | 1 | 2 | 0
Eye Pain (Eye disorders) | 0 | 1 | 2 | 0
Visual Acuity Reduced (Eye disorders) | 2 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 3 | 1 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Chills (General disorders) | 1 | 0 | 0 | 2
Gait Disturbance (General disorders) | 1 | 3 | 0 | 1
Oedema (General disorders) | 1 | 3 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 2
Eye Infection (Infections and infestations) | 1 | 0 | 2 | 0
Fungal Skin Infection (Infections and infestations) | 2 | 1 | 1 | 0
Helicobacter Infection (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 4 | 1 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 0 | 1 | 1
Haemorrhage Urinary Tract (Renal and urinary disorders) | 3 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 3 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 3 | 0 | 0
Urethral Pain (Renal and urinary disorders) | 2 | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 3 | 3 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 1
Nail Bed Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
These results are up to clinical cutoff (CCO) date 31 March 2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.